CLINICAL TRIAL: NCT03145844
Title: Evaluation of Efficacy and Safety of Direct Acting Agents in Hepatitis C Patients
Brief Title: Direct Acting Agents in Hepatitis C Patients
Acronym: HEPCTURKEY
Status: Completed | Type: Observational
Sponsor: Fehmi Tabak (Other)
Collaborators: Viral Hepatitis Society (Other)
Responsible Party: Sponsor-Investigator, Fehmi Tabak, Prof. Fehmi Tabak, Viral Hepatitis Society
Organization: Viral Hepatitis Society (Other)
Other Study IDs: HEPCTURKEY
Record Dates: First submitted 2017-05-03; First posted 2017-05-09 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Hepatitis C; Hepatitis C Relapse; Hepatitis C Recurrent
Keywords: DAA; Hepatitis
MeSH Terms: conditions — Hepatitis C; Hepatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Direct Acting Agents: No Intervention

SUMMARY:
This study is a retrospective study conducted at 36 sites. Planned target patient number is 1000.

DETAILED DESCRIPTION:
Approximately 36 centers will be included in Turkey. Centers will be selected from clinics of infection and clinical microbiology. The inclusion of 1000 patients was targeted. All data will be retrospectively collected from the medical records of the patients. Patient visit is not necessary.

ELIGIBILITY:
Inclusion Criteria:

* Patients who used direct acting agents for Hepatitis C

Exclusion Criteria:

* Patients younger then 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed as Hepatitis C and used direct acting agents.
Sampling Method: Non-Probability Sample
Enrollment: 2700 (Actual)
Dates: Start 2017-04-09 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Disease management with direct acting agents | Beginning of treatment - 12 weeks after the treatment ended (36 weeks)
  To assess disease management of chronic hepatitis C patients using direct acting agents (DAA) at national level, especially change in HCVRNA levels 12 weeks after the 24 weeks treatment (SVR12)

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Up to 48 weeks
  Adverse event list according to CTCAE v.4.03

CONTACTS AND LOCATIONS:
Overall Officials: Fehmi Tabak, Prof, Principal Investigator — Viral Hepatitis Society; Tansu Yamazhan, Prof, Study Director — Viral Hepatitis Society
Locations (1):
- Cerrahpasa Medical Faculty, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dirican E, Bal T, Onlen Y, Sarigul F, User U, Sari ND, Kurtaran B, Senates E, Gunduz A, Zerdali E, Karsen H, Batirel A, Karaali R, Guner HR, Yamazhan T, Kose S, Erben N, Ince NK, Koksal I, Oztoprak N, Yoruk G, Komur S, Kaya SY, Bozkurt I, Gunal O, Yildiz IE, Inan D, Barut S, Namiduru M, Tosun S, Turker K, Sener A, Hizel K, Baykam N, Duygu F, Bodur H, Can G, Gul HC, Tartar AS, Celebi G, Sunnetcioglu M, Karabay O, Kumbasar Karaosmanoglu H, Sirmatel F, Tabak OF. Assisting the Diagnosis of Cirrhosis in Chronic Hepatitis C Patients Based on Machine Learning Algorithms: A Novel Non-Invasive Approach. J Clin Lab Anal. 2025 Jun;39(12):e70054. doi: 10.1002/jcla.70054. Epub 2025 May 19. PMID 40384539